CLINICAL TRIAL: NCT06600594
Title: The Effect of Dance Training on Psychomotor Skills, Balance and Body Posture Control in Young Adults - the Involvement of Neurotrophic Factors
Brief Title: The Effect of Dance Training on Psychomotor, Biomechanical and Biochemical Parameters in Adults
Acronym: Dance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: SKE01-29/2022
Record Dates: First submitted 2024-02-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Psychomotor Status; Muscle Strain, Lower Leg; Muscle Strain Back; Balanced
Keywords: Dance Training; myometrics; blood tests; Balance; Psychomotor skills
MeSH Terms: conditions — Status Epilepticus; Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- KT - Control Group (No Intervention): Cosmetology and physiotherapy students who do not practice any sports
- PT - Beginner Group (Experimental): Students joining the "Podlasie" Song and Dance Ensemble - beginners
  Interventions: Other: Beginners dance training
- DT - Experienced Group (Active Comparator): Young adults trained from the "Podlasie" team with approximately 2-3 years of experience.
  Interventions: Other: Experience dance training

INTERVENTIONS:
Other: Beginners dance training — Trainings will be conducted twice a week for two hours. The training includes a general warm-up, polishing the steps, including regional dances, and then dancing entire dance routines.
  Arms: PT - Beginner Group
Other: Experience dance training — Trainings will be conducted twice a week for two hours. The training includes a general warm-up, polishing the steps, including regional dances, and then dancing entire dance routines.
  Arms: DT - Experienced Group

SUMMARY:
Clinical Trial, repeated-measures design, pilot study.

81 young adults, male (30) and female (51) underwent research protocol.

The aim of the research will be to assess the impact of long-term dance training on psychomotor performance, balance, body posture control and the level of neurotrophic factors in the blood in young adults.

People qualified for the study were divided into 3 groups depending on their dance experience:

1. KT young adults who do not exercise - cosmetology and physiotherapy students who do not practice any sports;
2. PT young adults - students joining the "Podlasie" Song and Dance Ensemble - beginners;
3. DT young adults trained from the "Podlasie" team with approximately 2-3 years of experience.

The DT group consisted 32 people (13 males and 19 females). In the beginners (PT) group were 25 people(6 males and 19 females) and 28(11 males and 17 females)were in KT group. DT and KT group were test one time (at the beginning) but the PT group was test 3 times ( at the beginning, 6 and 12 months later).

All groups have been subjected to comprehensive tests like anthropometric data, assessment of muscle strength, testing the biomechanical properties of the muscles of the lower and upper limbs and the shoulder girdle, testing postural stability in static and dynamic conditions, assessment of psychomotor skills, manual dexterity/ambidextrous and cognitive functions.

DETAILED DESCRIPTION:
I. The specific objectives were to investigate whether the dance training effect on:

1. Body composition
2. myometric variables (stiffness, flexibility and tension) of the muscle (trapezius upper part, quadriceps femoris, gastrocnemius muscle, patellar ligament proper)
3. concentration of selected biochemical factors (testosterone, brain-derived neurotrophic factor (BDNF)
4. muscle strength (flex and straighten the knee joint muscles)
5. postural stability ( dynamic and static conditions)
6. psychomotor skills (Simple reaction, Complex reaction, Eye-hand coordination, Spatial orientation)
7. manual dexterity/ambidextrous (Test Purdue Pegboard)
8. cognitive functions (TrailMaking Test (TMT) Parts A & B i STROOP 5.1 (ST))

II. Hypothese Dance as a form of long-term training improves psychomotor performance, balance and body posture control, as well as the level of neurotrophic factors in the blood in young adults.

III. Research Questions/Problems How will dance as a form of long-term training affect the psychomotor performance, balance and posture control of young adults? How can dancing as a form of long-term training change the properties (stiffness, flexibility, tension) of muscles at rest and the strength of the muscles of the lower and upper limbs and the shoulder girdle in young adults? How does dancing as a form of long-term training affect the level of neurotrophic factors and androgen hormones in the blood in young adults? Is there a correlation between the level of BDNF and testosterone in the blood and psychomotor performance, balance, body posture control, properties (stiffness, elasticity, tension) and strength of selected muscles in young adults after a dance training process? Does a 12-month dance training process cause similar changes in psychomotor efficiency, balance and body posture control as a 6-month training process in young adults?

IV. The course of the research Before and during the intervention cycle, the dancers were subjected to biomechanical and biochemical tests. Fasting blood was collected on the day of the examination to determine biochemical parameters. Before starting the study, patients completed a research consent form and an abbreviated version of the Minnesota Physical Activity Test (IPQ). During each cycle of tests, myometric measurements of muscle tension, stiffness and elasticity were performed using the Myoton Pro 3 device (Tallinn, Estonia), assessment of muscle strength using the Biodex System 4-ORO, postural stability in static and dynamic conditions using the Accusway Plus AMTI posturographic plate, assessment of psychomotor skills using a computer program, assessment of two-handed manual dexterity (Purdue Pegboard Test) and cognitive functions (TrailMaking Tesr (TMT) Parts A & B and STROOP 5.1 (ST). The research was conducted in 3 stages: at the beginning, after 6 months and after 12 months after introducing dance training.

V. Research Methods

1. Anthropometric data - Body composition analysis will be performed using the Tanita BC 418 ma electronic system (Tanita Corporation, Tokyo, Japan T174) device to determine body weight, fat content and skeletal muscle mass. The height of the subjects will be measured. The BMI index will be determined based on body weight and height using the formula BMI = body weight [kg] / (body height [m])2 The following measurement methods will be used to measure muscle properties and strength
2. Assessment of muscle strength - Muscle strength will be assessed using Biodex System 4-PRO - an isokinetic dynamometer: Before starting the measurements, the subjects perform a 5-minute warm-up on a cycle ergometer. Then they take a standard position on the chair and are stabilized with belts in the manner recommended by the device manufacturer. The range of motion in the joint is limited to 90 degrees. To assess the torque of the muscles that flex and straighten the limb in the knee joint, an isokinetic test will be used, performed at two constant, commonly used angular velocities of the lower leg: 60 deg/s and 180 deg/s. The test consists of a series of 5 straightening and bending movements at a lower speed and 10 movements at a higher speed, preceded in both cases by three trials, which are performed with moderate muscle involvement. During the measurements, the moments of muscle forces of the knee flexors and extensors will be recorded and saved in the form of text files. Additionally, the following values will be read from the measurement protocol of each subject for both angular velocities:

   * maximum moment of force of the muscles that extend (Mpk) and bend (Mzk) the knee joint;
   * relative moment of the maximum force of the muscles that extend and bend the knee joint (the maximum moment of the muscles that extend (Mpk) and flexion (Mzk) the knee joint is determined by the body weight of the examined person)
3. Testing the biomechanical properties of the muscles of the lower and upper limbs and the shoulder girdle (stiffness, elasticity, tension) at rest using the Myoton PRO myometer (Estonia) The muscle properties were tested using a Myoton Pro 3 miometer (Myoton, Tallinn, Estonia). The measurement is non-invasive and fast, it takes from 3 to 30 seconds depending on the selected option. In the presented work, the 10 measurement repetition mode was selected, from which the device software calculated the average for each of the three parameters (tension, stiffness and elasticity) and saved it in the device memory. The measurement consisted in placing the measuring tip of the myometer always perpendicular to the skin surface at a strictly defined point. The researcher moved the device towards the examined tissue until the green light on the body of the device turned on. Such an operation activates the electromagnetic mechanism, which generated mechanical impulses with a constant force deforming the muscle at the measuring point through the moved measuring tip. The meter automatically performed a series of pulses (10), and the researcher held the device steadily in the selected position. The pressure of the tip (punch) is short (10 ms) and of low force (0.40 N), which does not cause a neurological reflex muscle contraction response. The impulse caused mechanical vibrations of the examined muscle, according to which the following parameters were calculated after automatic processing by the accelerometric recording processor:

   * F (frequency) - it determines the muscle tension and is calculated as the maximum frequency from the power of the accelerometric signal spectrum and is expressed as in hertz [Hz].
   * S (stiffness) - is calculated from the formula S-MYO = amax. mprobe / ^ l, where amax is the maximum acceleration of the striking measuring tip [kg], a ^ l is the maximum distance the stylus has moved [m]. This parameter is expressed in [N / m] and determines the force generated by the measuring tip of the myometer needed to deform the tested tissue to a specific depth.
   * D (decrement) - free decrease of vibration calculated from the logarithm.
4. Postural stability testing in static and dynamic conditions - will be performed using the AccuSway Plus AMTI postural plate. The test of postural stability in static conditions will be expressed by the characteristics of the swaying of the center of pressure of the feet on the ground recorded in a standing position (as calm as possible) for 30 seconds. under eyes open [OO] and eyes closed [OZ] conditions. An attempt will be made to measure postural stability in static conditions with a simultaneous cognitive task (reading text or counting). The test of postural stability in dynamic conditions will be determined by the limit of stability [Limit of stability - LOS [cm] expressed by testing the maximum forward and backward body tilt in OO and OZ conditions. The subjects will be asked to keep their body stiffened, bend as far as possible in the anterior and posterior direction - AP-LOS, and then maintain each extreme position for 2 s. The entire plantar surface of the feet should be in contact with the ground at all times.

   The following methods will be used to assess psychomotor skills:
5. Assessment of psychomotor skills - To assess selected elements of psychomotor skills, a computer program will be used, which is part of a set of computer tests of coordination abilities.

The following tests will be used in the research:

* Simple reaction - measurement of simple reaction time to a visual stimulus. In measuring the simple reaction time, I will use the arrhythmic emission of 11 impulses appearing on the monitor. The shorter the test time, the better the result.
* Complex reaction - measurement of complex reaction time to visual stimuli. In measuring simple reaction time, arrhythmic emission of 11 impulses will be used - Assessment of the level of selected fitness elements. 121 words appearing on the monitor. The shorter the test time, the better the result.
* Eye-hand coordination - the effect of eye-hand coordination will be measured using the arrhythmic emission of 42 impulses appearing on the monitor. The shorter the test time, the better the result.
* Spatial orientation - the measurement of the effect of orientation and perception will be analyzed using 4 levels of difficulty. The measure of assessing the level of spatial orientation will be the percentage of correctness of the test task performance (spatial orientation index). The higher the percentage obtained in the sample, the better the test result.

  9. Blood collection, measurements and hematological parameters In the study groups, blood samples for measurement of blood variables will be collected from the basilic vein at rest in the morning between 8:00 a.m. and 10:00 a.m. on an empty stomach. Blood for serum measurements will be collected in anticoagulant-free tubes with coagulation activator centrifuged at 653 × g for 10 minutes at 4°C. The serum will be stored at -80°C for further analysis. Total and differential blood counts will be analyzed using standard hematology procedures on the ADVIA 60 model analyzer.

  10. Measurements of biochemical markers in serum We will assess the level of BDNF testosterone in the serum using an enzyme-linked immunosorbent assay (ELISA) and molecular biology techniques. The serum will be tested for BDNF, testosterone, using an enzyme-linked immunosorbent assay (ELISA) kit after appropriate dilution with the block and sample solution (provided in the kit). A microplate reader (BioTek, Biokom, USA) set at 450 nm will be used to determine the values of neurotrophic factors, testosterone and cytokine levels.

VI. Statistical analysis The obtained results will be presented as the arithmetic mean ± mean arithmetic error (SEM) from n independent measurements. The statistical analysis will be performed in the STATISTICA v. 10 program. The Shapiro-Wilk test will be used to check the normality of the distribution of concentrations of biochemical factors in the serum, biomechanical parameters, muscle properties parameters, myometric tests, body balance muscle strength and psychomotor skills. When significant deviations from normal distribution were demonstrated, further analyzes were performed using non-parametric tests. In the case of analysis of comparisons of several measurements (more than two), Friedman's ANOVA will be used, and when there are differences between variables, the Post-Hoc For Friedman test will be used. In the comparative analysis of two measurements, a non-parametric test for two dependent samples will be used: Wilcoxon pairwise order. A correlation analysis (Pearson or Spearman correlation coefficient) will be performed between the data of biochemical markers (BDNF, testosterone) and biomechanical results, muscle properties and psychomotor performance parameters. The results will be considered statistically significant at the significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* age
* preferring dance as a form of exercise

Exclusion Criteria:

* age under 19 or older than 25
* any chronic diseases
* any diseases
* practicing sports professionally for PT group

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Stiffness | Myometric measurements were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training
  S (stiffness) - is calculated from the formula S-MYO = amax. mprobe / ^ l, where amax is the maximum acceleration of the striking measuring tip [kg], a ^ l is the maximum distance the stylus has moved [m]. This parameter is expressed in [N / m] and determines the force generated by the measuring tip of the myometer needed to deform the tested tissue to a specific depth
Muscle Elasticity | Myometric measurements were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training
  D (decrement) - free decrease of vibration calculated from the logarithm
Blood parameters | [Time Frame: Peripheral blood from the antecubital vein was collected on an empty stomach between 6:00 a.m. and 9:00 a.m. before each examination (at baseline, 6 months and 12 months after the start of the intervention)]
  The concentration of androgen factors, testosterone and BNDF (brain-derived neurotrophic factor) was determined using the immunochemical ELISA method in accordance with the kit manufacturer's instructions (R&D systems, London UK).
Muscle Tension | Myometric measurements were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training
  F (frequency) - it determines the muscle tension and is calculated as the maximum frequency from the power of the accelerometric signal spectrum and is expressed as in hertz [Hz].

SECONDARY OUTCOMES:
Maximum torque of the muscles that extend (Mpk) and flexion (Mzk) the knee joint | Muscle strength was performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  To assess the torque of the muscles that flex and extend the limb in the knee joint, an isokinetic test will be used, performed at two constant, commonly used angular velocities of the lower leg: 60 deg/s and 180 deg/s.
Relative moment of the maximum force of the muscles that extend and bend the knee joint (maximum moment of the muscles that extend (Mpk) and flexing (Mzk) knee joint is determined by the body weight of the examined person | Muscle strength was performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  To assess the torque of the muscles that flex and extend the limb in the knee joint, an isokinetic test will be used, performed at two constant, commonly used angular velocities of the lower leg: 60 deg/s and 180 deg/s.
Dynamic and static postural stability | Balance was performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  The test of postural stability in static conditions will be expressed by the characteristics of the swaying of the center of pressure of the feet on the ground recorded in a standing position (as calm as possible) for 30 seconds. under eyes open [OO] and eyes closed [OZ] conditions.
Simple reaction | Psychomotor skills were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  Measurement of simple reaction time to a visual stimulus. In measuring the simple reaction time, I will use the arrhythmic emission of 11 impulses appearing on the monitor. The shorter the test time, the better the result.
Complex reaction | Psychomotor skills were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  Measurement of complex reaction time to visual stimuli. In measuring simple reaction time, arrhythmic emission of 11 impulses will be used - Assessment of the level of selected fitness elements. 121 words appearing on the monitor. The shorter the test time, the better the result.
Eye-hand coordination | Psychomotor skills were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  To measure the effect of eye-hand coordination, the arrhythmic emission of 42 impulses appearing on the monitor will be used. The shorter the test time, the better the result.
Spatial orientation | Psychomotor skills were performed once in the DT and KT groups. However, in the PT group, the study was carried out 3 times, at the beginning, after 6 months and 12 months after the start of dance training.
  The measurement of the orientation and perception effect will be analyzed using 4 levels of difficulty. The measure of assessing the level of spatial orientation will be the percentage of correctness of the test task performance (spatial orientation index). The higher the percentage obtained in the sample, the better the test result.

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Łuć, Study Director — Regional Research and Development Center in Biała Podlaska
Locations (1):
- Regional Research and Development Center, Biała Podlaska, Bialski, Poland

IPD SHARING:
Plan to Share IPD: No